CLINICAL TRIAL: NCT01956357
Title: Chronic Effects of Two Aerobic-training Models Performed in Water and on Dry Land in Patients With Type 2 Diabetes Mellitus (T2DM).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Rodrigo Sudatti Delevatti, Effects of two models of aerobic training performed in different environments in patients with type 2 diabetes mellitus, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 54475
Record Dates: First submitted 2013-09-27; First posted 2013-10-08 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: aquatic exercises;; deep water running;; diabetes;; blood glucose;; inflammation.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Inflammation | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Aquatic exercise (Experimental): The aquatic aerobic training had a duration of 12 weeks and adopted the interval-training method, with intensities ranging between 85 and 100% of second ventilatory threshold (VT2) and total duration of 45 minute per session.
  The sessions consisted of warm up, main part and calm down. The warm-up consisted of a walk in deep water at low intensity for three minutes. The main part was intended to aerobic training in deep water, in which subjects walked and / or ran, depending on your fitness level found in pre-training test. The calm down consisted of walking in deep water at low intensity for two minutes and stretching standardized, emphasizing the muscles worked in the main part of the session, with a total duration of approximately five minutes.
  Interventions: Other: Aquatic exercise
- Land exercise (Experimental): The land aerobic training had a duration of 12 weeks and adopted the interval-training method, with intensities ranging between 85 and 100% of second ventilatory threshold (VT2) and total duration of 45 minute per session.
  The sessions consisted of warm up, main part and calm down. The warm-up consisted of a walk in athletic track at low intensity for three minutes. The main part was intended to aerobic training in athletic track, in which subjects walked and / or ran, depending on your fitness level found in pre-training test. The calm down consisted of walking in athletic track at low intensity for two minutes and stretching standardized, emphasizing the muscles worked in the main part of the session, with a total duration of approximately five minutes.
  Interventions: Other: Land Exercise

INTERVENTIONS:
Other: Aquatic exercise
  Arms: Aquatic exercise
Other: Land Exercise
  Arms: Land exercise

SUMMARY:
The aim of this study was to analyse the acute and chronic effects of two aerobic-training models performed in water and on dry land on cardiorespiratory, functional, metabolic, hormonal and quality-of-life parameters in patients with type 2 diabetes mellitus (T2DM).

ELIGIBILITY:
Inclusion Criteria:

The clinical diagnosis of type 2 diabetes mellitus. Not be performing regular and systematic physical exercise for at least three months.

Exclusion Criteria:

Uncontrolled hypertension. Autonomic neuropathy. Severe peripheral neuropathy. Proliferative diabetic retinopathy. Severe nonproliferative diabetic retinopathy. Uncompensated heart failure. Peripheral amputations. Chronic renal failure (GFR by MDRD <30). Muscle or joint injury that prevents physical exercises.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | Baseline and after 12 weeks of intervention

SECONDARY OUTCOMES:
Fasting plasma glucose. | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Postprandial glucose | Baseline and after 12 weeks of intervention.
Fasting insulin. | Baseline and after 12 weeks of intervention.
Insulin resistance (HOMA-IR). | Baseline and after 12 weeks of intervention.
Total cholesterol. | Baseline and after 12 weeks of intervention.
High density lipoprotein. | Baseline and after 12 weeks of intervention.
Low density lipoprotein. | Baseline and after 12 weeks of intervention.
Triglycerides. | Baseline and after 12 weeks of intervention.
Plasma renin activity. | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Angiotensin II. | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
C-reactive protein ultrasensitive. | Baseline and after 12 weeks of intervention.
8-isoprostane | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Content of reative species (DCF) | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Water-soluble Fluorescent Substances | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Oxidation of tyrosine residues | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Oxidation of tryptophan | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
superoxide dismutase (SOD) | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Catalase (CAT) | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Glutathione peroxidase (GPX) | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Total radical-trapping antioxidant potential (TRAP) | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Interleukin 1β | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Interleukin 10 | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Leukocyte DNA Methylation | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Purines | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Interleukin 6 | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.
Global Histone Deacetylases activity | Before and after a session of 45 minutes of exercise; baseline and after 12 weeks of intervention.

OTHER OUTCOMES:
Peak oxygen consumption. | Baseline and after 12 weeks of intervention.
Timed up and go in habitual speed and maximal speed. | Baseline and after 12 weeks of intervention.
Oxygen uptake at ventilatory threshold. | Baseline and after 12 weeks of intervention.
Percentage of oxygen consumption at ventilatory threshold. | Baseline and after 12 weeks of intervention.
Systolic blood pressure. | Baseline and after 12 weeks of intervention.
Diastolic blood pressure | Baseline and after 12 weeks of intervention.
Resting heart rate. | Baseline and after 12 weeks of intervention.
Quality of life. | Baseline and after 12 weeks of intervention.
Depressive symptoms. | Baseline and after 12 weeks of intervention.
Sleep quality. | Baseline and after 12 weeks of intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo S Delevatti, MSc, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Physical Education School of Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande Do Sil, Brazil

REFERENCES:
- [Derived] S Delevatti R, Schuch FB, Kanitz AC, Alberton CL, Marson EC, Lisboa SC, Pinho CDF, Bregagnol LP, Becker MT, Kruel LFM. Quality of life and sleep quality are similarly improved after aquatic or dry-land aerobic training in patients with type 2 diabetes: A randomized clinical trial. J Sci Med Sport. 2018 May;21(5):483-488. doi: 10.1016/j.jsams.2017.08.024. Epub 2017 Sep 6. PMID 28935128
- [Derived] Delevatti RS, Pinho CD, Kanitz AC, Alberton CL, Marson EC, Bregagnol LP, Lisboa SC, Schaan BD, Kruel LF. Glycemic reductions following water- and land-based exercise in patients with type 2 diabetes mellitus. Complement Ther Clin Pract. 2016 Aug;24:73-7. doi: 10.1016/j.ctcp.2016.05.008. Epub 2016 May 10. PMID 27502804